CLINICAL TRIAL: NCT02625155
Title: Standard of Care Versus Urine Testing With Selective PHarmacogenomics for Effective Drug and Dosing REgimens: SPHERE
Brief Title: Standard of Care Versus Urine Testing With Selective PHarmacogenomics for Effective Drug and Dosing REgimens
Acronym: SPHERE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: InSource Diagnostics (Industry)
Collaborators: Syntactx (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-001
Record Dates: First submitted 2015-11-25; First posted 2015-12-09 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2017-03

CONDITIONS: Target Drug-related Adverse Events
Keywords: Pharmacogenomics; Urine Drug Testing; antidepressants; benzodiazepines; opioids; muscle relaxants; non-steroidal anti-inflammatory agents; TDRAE
MeSH Terms: conditions — Muscle Hypotonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (SOC Arm) (Other): Standard of Care UDT
  Interventions: Other: Urine diagnostic testing as SOC, drug regimen changes per SOC
- Selective PGx Testing (Test Arm) (Other): Standard of Care UDT with selective PGx testing
  Interventions: Other: Urine diagnostic testing with selective PGx testing, drug regimen changes based on PGx test results

INTERVENTIONS:
Other: Urine diagnostic testing as SOC, drug regimen changes per SOC
  Arms: Standard of Care (SOC Arm)
Other: Urine diagnostic testing with selective PGx testing, drug regimen changes based on PGx test results
  Arms: Selective PGx Testing (Test Arm)

SUMMARY:
The purpose of this study is to determine whether the addition of selective pharmacogenomic (PGx) testing as determined by Urine Drug Testing (UDT) adds a clinical benefit as evidenced by a reduction in Target Drug-related Adverse Events (TDRAE) over the period following enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 12 years of age or older;
2. Subject or legal representative is able and willing to provide informed consent;
3. Subject has had a TDRAE including ineffective therapeutic response within the last 60 days or is a new patient to the treating healthcare provider's practice;
4. Subject is scheduled for or is planned to be scheduled for UDT, ordered as per the treating healthcare provider's local standard of care;
5. Subject is currently receiving or the subject's treating healthcare provider is considering treatment with at least one target drug listed below and metabolized by one or more genes considered in this study: Amitriptyline, Imipramine, Diazepam, Alprazolam, Codeine, Hydrocodone, Oxycodone, Methadone, Meperidine, Fentanyl and Carisoprodol.

Exclusion Criteria:

1. Prior history of PGx testing for genes specific to any of the target drugs in the past;
2. PGx testing is deemed mandatory in the opinion of the treating healthcare provider;
3. History of liver or renal transplantation;
4. Receiving chronic hemodialysis or peritoneal dialysis;
5. Currently hospitalized or in a long-term care facility;
6. Participation in another clinical trial that would, in the Investigator's opinion, interfere with the conduct of this study;
7. Subject or subject's guardian or advocate is unable to provide an accurate history of the subject's medical history, medications, and symptoms.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 14000 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects who experience target drug-related adverse events (TDRAE) over the 90-day period following enrollment | 90 days

SECONDARY OUTCOMES:
All TDRAE as quantified within each of the four classes of medications | 90 days
TDRAE driving a change in the subject's drug regimen (dose change, discontinuation, substation, or addition of a new drug) | 90 days
Severe TDRAE, defined as a TDRAE that meets the criteria for a Serious Adverse Event | 90 days
Ineffective therapeutic response, determined by the Investigator | 90 days
Supra-therapeutic response, as determined by the Investigator | 90 days
Frequency of subjects with changes in drug regimen | 90 days
Healthcare resource utilization, as measured by the number of outpatient clinic visits, emergency room/urgent care visits, and hospitalizations; tabulated over the 90-day period following enrollment | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Donald H. Deaton, Jr., DO, Tazewell, Tennessee, United States

REFERENCES:
- [Background] Phimister EG, Feero WG, Guttmacher AE. Realizing genomic medicine. N Engl J Med. 2012 Feb 23;366(8):757-9. doi: 10.1056/NEJMe1200749. No abstract available. PMID 22356329
- [Background] Rebsamen MC, Desmeules J, Daali Y, Chiappe A, Diemand A, Rey C, Chabert J, Dayer P, Hochstrasser D, Rossier MF. The AmpliChip CYP450 test: cytochrome P450 2D6 genotype assessment and phenotype prediction. Pharmacogenomics J. 2009 Feb;9(1):34-41. doi: 10.1038/tpj.2008.7. Epub 2008 Jul 1. PMID 18591960
- [Background] Hicks JK, Bishop JR, Sangkuhl K, Muller DJ, Ji Y, Leckband SG, Leeder JS, Graham RL, Chiulli DL, LLerena A, Skaar TC, Scott SA, Stingl JC, Klein TE, Caudle KE, Gaedigk A; Clinical Pharmacogenetics Implementation Consortium. Clinical Pharmacogenetics Implementation Consortium (CPIC) Guideline for CYP2D6 and CYP2C19 Genotypes and Dosing of Selective Serotonin Reuptake Inhibitors. Clin Pharmacol Ther. 2015 Aug;98(2):127-34. doi: 10.1002/cpt.147. Epub 2015 Jun 29. PMID 25974703
- [Background] Crews KR, Gaedigk A, Dunnenberger HM, Klein TE, Shen DD, Callaghan JT, Kharasch ED, Skaar TC; Clinical Pharmacogenetics Implementation Consortium. Clinical Pharmacogenetics Implementation Consortium (CPIC) guidelines for codeine therapy in the context of cytochrome P450 2D6 (CYP2D6) genotype. Clin Pharmacol Ther. 2012 Feb;91(2):321-6. doi: 10.1038/clpt.2011.287. Epub 2011 Dec 28. PMID 22205192
- [Background] Sohn DR, Kusaka M, Ishizaki T, Shin SG, Jang IJ, Shin JG, Chiba K. Incidence of S-mephenytoin hydroxylation deficiency in a Korean population and the interphenotypic differences in diazepam pharmacokinetics. Clin Pharmacol Ther. 1992 Aug;52(2):160-9. doi: 10.1038/clpt.1992.125. PMID 1505151
- [Background] Bernard S, Neville KA, Nguyen AT, Flockhart DA. Interethnic differences in genetic polymorphisms of CYP2D6 in the U.S. population: clinical implications. Oncologist. 2006 Feb;11(2):126-35. doi: 10.1634/theoncologist.11-2-126. PMID 16476833
- [Background] Wijnen PA, Op den Buijsch RA, Drent M, Kuijpers PM, Neef C, Bast A, Bekers O, Koek GH. Review article: The prevalence and clinical relevance of cytochrome P450 polymorphisms. Aliment Pharmacol Ther. 2007 Dec;26 Suppl 2:211-9. doi: 10.1111/j.1365-2036.2007.03490.x. PMID 18081664
- [Background] Linares OA, Fudin J, Daly AL, Boston RC. Individualized Hydrocodone Therapy Based on Phenotype, Pharmacogenetics, and Pharmacokinetic Dosing. Clin J Pain. 2015 Dec;31(12):1026-35. doi: 10.1097/AJP.0000000000000214. PMID 25621429
- [Background] Falzone E, Hoffmann C, Keita H. Postoperative analgesia in elderly patients. Drugs Aging. 2013 Feb;30(2):81-90. doi: 10.1007/s40266-012-0047-7. PMID 23288604
- [Background] Balhara YP, Jain R. A urinalysis-based study of buprenorphine and non-prescription opioid use among patients on buprenorphine maintenance. J Pharmacol Pharmacother. 2012 Jan;3(1):15-9. doi: 10.4103/0976-500X.92496. PMID 22368411
- [Background] Christo PJ, Manchikanti L, Ruan X, Bottros M, Hansen H, Solanki DR, Jordan AE, Colson J. Urine drug testing in chronic pain. Pain Physician. 2011 Mar-Apr;14(2):123-43. PMID 21412368
- [Background] Uher R, Farmer A, Henigsberg N, Rietschel M, Mors O, Maier W, Kozel D, Hauser J, Souery D, Placentino A, Strohmaier J, Perroud N, Zobel A, Rajewska-Rager A, Dernovsek MZ, Larsen ER, Kalember P, Giovannini C, Barreto M, McGuffin P, Aitchison KJ. Adverse reactions to antidepressants. Br J Psychiatry. 2009 Sep;195(3):202-10. doi: 10.1192/bjp.bp.108.061960. PMID 19721108
- [Background] Vilhelmsson A, Svensson T, Meeuwisse A, Carlsten A. What can we learn from consumer reports on psychiatric adverse drug reactions with antidepressant medication? Experiences from reports to a consumer association. BMC Clin Pharmacol. 2011 Oct 25;11:16. doi: 10.1186/1472-6904-11-16. PMID 22026961
- [Background] Fabbri C, Serretti A. Pharmacogenetics of major depressive disorder: top genes and pathways toward clinical applications. Curr Psychiatry Rep. 2015 Jul;17(7):50. doi: 10.1007/s11920-015-0594-9. PMID 25980509
- [Background] Kreyenbuhl JA, Valenstein M, McCarthy JF, Ganoczy D, Blow FC. Long-term antipsychotic polypharmacy in the VA health system: patient characteristics and treatment patterns. Psychiatr Serv. 2007 Apr;58(4):489-95. doi: 10.1176/ps.2007.58.4.489. PMID 17412850
- [Background] Gurwitz JH, Field TS, Avorn J, McCormick D, Jain S, Eckler M, Benser M, Edmondson AC, Bates DW. Incidence and preventability of adverse drug events in nursing homes. Am J Med. 2000 Aug 1;109(2):87-94. doi: 10.1016/s0002-9343(00)00451-4. PMID 10967148
- [Background] Moeller KE, Lee KC, Kissack JC. Urine drug screening: practical guide for clinicians. Mayo Clin Proc. 2008 Jan;83(1):66-76. doi: 10.4065/83.1.66. PMID 18174009
- [Background] Crews KR, Hicks JK, Pui CH, Relling MV, Evans WE. Pharmacogenomics and individualized medicine: translating science into practice. Clin Pharmacol Ther. 2012 Oct;92(4):467-75. doi: 10.1038/clpt.2012.120. Epub 2012 Sep 5. PMID 22948889
- [Background] Hamburg MA, Collins FS. The path to personalized medicine. N Engl J Med. 2010 Jul 22;363(4):301-4. doi: 10.1056/NEJMp1006304. Epub 2010 Jun 15. No abstract available. PMID 20551152
- [Background] Yiannakopoulou E. Pharmacogenomics and Opioid Analgesics: Clinical Implications. Int J Genomics. 2015;2015:368979. doi: 10.1155/2015/368979. Epub 2015 May 14. PMID 26075211
- [Background] Stanek EJ, Sanders CL, Taber KA, Khalid M, Patel A, Verbrugge RR, Agatep BC, Aubert RE, Epstein RS, Frueh FW. Adoption of pharmacogenomic testing by US physicians: results of a nationwide survey. Clin Pharmacol Ther. 2012 Mar;91(3):450-8. doi: 10.1038/clpt.2011.306. Epub 2012 Jan 25. PMID 22278335
- [Background] Deverka PA. Pharmacogenomics, evidence, and the role of payers. Public Health Genomics. 2009;12(3):149-57. doi: 10.1159/000189627. Epub 2009 Feb 10. PMID 19204417
- [Background] Local Coverage Determination (LCD): CYP2C19, CYP2D6, CYP2C9, and VKORC1 Genetic Testing (L35472). 2015. (Accessed 8/10/2015, at https://www.cms.gov/medicare-coverage-database/details/lcd-details.aspx?LCDId=35472&ContrId=357.)
- [Background] Manchikanti L, Atluri S, Trescot AM, Giordano J. Monitoring opioid adherence in chronic pain patients: tools, techniques, and utility. Pain Physician. 2008 Mar;11(2 Suppl):S155-80. PMID 18443638
- [Background] Konstantinova SV, Normann PT, Arnestad M, Karinen R, Christophersen AS, Morland J. Morphine to codeine concentration ratio in blood and urine as a marker of illicit heroin use in forensic autopsy samples. Forensic Sci Int. 2012 Apr 10;217(1-3):216-21. doi: 10.1016/j.forsciint.2011.11.007. Epub 2011 Dec 2. PMID 22137531
- [Background] Standridge JB, Adams SM, Zotos AP. Urine drug screening: a valuable office procedure. Am Fam Physician. 2010 Mar 1;81(5):635-40. PMID 20187600
- [Background] Disability Evaluation Under Social Security. (Accessed 3/5/2014, 2014, at http://www.ssa.gov/disability/professionals/bluebook/general-info.htm.)
- [Background] Inter-agency guideline for opioid dosing for chronic non-cancer pain.2010.
- [Background] National Bioeconomy Blueprint. The White House; 2012:48.
- [Background] World Guide for Drug Use and Pharmacogenomics. Corunna, Spain: EuroEspes Publishing; 2012.
- [Background] Model policy on the use of opioid analgesics in the treatment of chronic pain. Federation of State Medical Boards; 2013.
- [Background] ACOEM. Guidelines for the Chronic Use of Opioids. 2 ed: American College of Occupational and Environmental Medicine.
- [Background] Michna E, Jamison RN, Pham LD, Ross EL, Janfaza D, Nedeljkovic SS, Narang S, Palombi D, Wasan AD. Urine toxicology screening among chronic pain patients on opioid therapy: frequency and predictability of abnormal findings. Clin J Pain. 2007 Feb;23(2):173-9. doi: 10.1097/AJP.0b013e31802b4f95. PMID 17237667
- [Background] Wiedemer NL, Harden PS, Arndt IO, Gallagher RM. The opioid renewal clinic: a primary care, managed approach to opioid therapy in chronic pain patients at risk for substance abuse. Pain Med. 2007 Oct-Nov;8(7):573-84. doi: 10.1111/j.1526-4637.2006.00254.x. PMID 17883742
- [Background] Gandhi TK, Weingart SN, Borus J, Seger AC, Peterson J, Burdick E, Seger DL, Shu K, Federico F, Leape LL, Bates DW. Adverse drug events in ambulatory care. N Engl J Med. 2003 Apr 17;348(16):1556-64. doi: 10.1056/NEJMsa020703. PMID 12700376
- [Background] Manchikanti L, Manchikanti KN, Pampati V, Cash KA. Prevalence of side effects of prolonged low or moderate dose opioid therapy with concomitant benzodiazepine and/or antidepressant therapy in chronic non-cancer pain. Pain Physician. 2009 Jan-Feb;12(1):259-67. PMID 19165308